CLINICAL TRIAL: NCT06530212
Title: Sleeve Gastrectomy With Jejuno-ieal Bypass
Brief Title: Sleeve Gastrectomy With Jejuno-ileal Bypass Versus Single Anastomosis Sleeve Jejunal Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, professor of general and bariatric surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ac.med.24.34
Record Dates: First submitted 2024-07-17; First posted 2024-07-31 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGJIB (Experimental)
  Interventions: Procedure: SGJIB
- SAS-JB (Active Comparator)
  Interventions: Procedure: SAS-JB

INTERVENTIONS:
Procedure: SGJIB — sleeve gastrectomy with jejunoileal bypass with anastomosis between the jejunum at about 100 cm from the duodeno-jejunal flexure and the ileum at 250 cm from the ileocaecal junction.
  Arms: SGJIB
Procedure: SAS-JB — single anastomosis sleeve jejunal bypass (SAS-JB) with biliary limb equal one third of total intestinal length.
  Arms: SAS-JB

SUMMARY:
sleeve gastrectomy with jejunoileal bypass (SGJIB) is a novel technique for the surgical treatment of obesity. The aim of the study is to compare this maneuver with single anastomosis sleeve jejunal bypass (SAS-JB)

DETAILED DESCRIPTION:
200 patients will be randomly divided into to equal . Group 1 will be operated by sleeve gastrectomy with jejunoileal bypass with the anastomosis between the jejunum at about 100 cm from the duodeno-jejunal flexure and the ileum at 250 cm from the ileocaecal junction. and group 2 will be operated by single anastomosis sleeve jejunal bypass (SAS-JB) with biliary limb equal one third of total intestinal length.

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Stoma complications | one year
  any complication due to sleeve jejunal anastomosis

SECONDARY OUTCOMES:
weight loss at one year | one year
  the effect of the 2 procedures on weight measured by percentage of excess weight loss
improvement of comorbidities | one year
  change in comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Sewefy, professor, Principal Investigator — Minia University, faculty of medicine; Taha Kayed, MD, Study Director — Minia University, faculty of medicine
Locations (1):
- Faculty of medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No